CLINICAL TRIAL: NCT02332512
Title: A Randomized, Double-blind, Placebo-controlled, Phase III Trial of Apatinib as 3rd/4th Line Treatment in Patients With Advanced Non-Squamous Non-Small Cell Lung Cancer Harboring Wild-type Epidermal Growth Factor Receptor (EGFR)
Brief Title: Study of Apatinib as 3rd/4th Line Treatment in Patients With Advanced Non-Squamous Non-small Cell Lung Cancer Harboring Wild-type Epidermal Growth Factor Receptor (EGFR)
Acronym: ANSWER
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR-APTN-Ⅲ-NSCLC-02
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Non-squamous non-small cell lung cancer; Wild-type EGFR; 3rd/4th line treatment; apatinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — apatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apatinib (Experimental): Apatinib tablet administered orally, 750 mg,once daily until progression
  Interventions: Drug: Apatinib
- Placebo (Placebo Comparator): Placebo tablet administered orally, once a day until progression
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apatinib
  Arms: Apatinib
Drug: Placebo
  Arms: Placebo

SUMMARY:
Apatinib is a new kind of selective Vascular Endothelial Growth Factor Receptor 2(VEGFR-2) tyrosine kinase inhibitor (TKI). The investigators have finished the preclinical,phase I and phase II clinical studies and found its promising anti-tumor activity and tolerable toxicities. A disease-control rate of 61.1% and a mPFS of 4.7 months were showed in apatinib phase II study in patients with NSCLC.

The study aims to compare the efficacy and safety of apatinib to placebo in advanced non-squamous non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects >/= 18 years and </=70 years of age at the time of Informed Consent.
2. Advanced relapsed or refractory predominantly NSCLC with documented wild-type EGFR.
3. At least one measurable lesion according to RECIST 1.1.
4. Failure of second line of chemotherapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Patients must have recovered from any AEs of prior treatments before randamization.
7. Adequate bone marrow,liver and renal function as assessed by the following laboratory tests conducted within 1 week before randomization. HB ≥ 90g/L; ANC≥1.5×10E+9/L; PLT≥80×10E+9/L; ALT and AST < 2.5×ULN; TBIL ≤1.25×ULN; Cr ≤1.25×ULN;CL>45 ml/min.
8. Life expectancy of at least three months.
9. Written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. Presence of types of small-cell, squamous-cell, adeno-squamous-cell lung cancer.
2. Pregnant or breast-feeding women.
3. Suffered from grade II or above myocardial ischemia or myocardial infarction, uncontrolled arrhythmias (including QT interval male ≥ 450 ms, female≥ 470 ms).Severe or uncontrolled systemic disease such as clinically significant hypertension(systolic pressure >/= 140 mm Hg and/or diastolic pressure >/= 90 mm Hg), and Grade III-IV cardiac insufficiency, according to NYHA criteria or echocardiography check: LVEF<50%.
4. Factors to affect oral administration(inability to swallow tablets,GI tract resection, chronic bacillary diarrhea and intestinal obstruction).
5. Coagulation disfunction,hemorrhagic tendency or receiving anticoagulant therapy>/= CTCAE 2 pneumorrhagia or >/= CTCAE 3 hemorrhage in other organs within 4 weeks.
6. Bone fracture or wounds that was not cured.
7. Arterial thrombus or phlebothrombosis within 12 months and taking anticoagulant agents.
8. Mental diseases and psychotropic substances abuse.
9. Previous treatment with an trial agent within 4 weeks
10. Previous treatment with VEGFR,platelet derived growth factor receptor(PDGFR) TKIs.
11. Proteinuria ≥ (++) or 24 hours total urine protein > 1.0 g.
12. Other coexisting malignant disease (except basal-cell carcinoma and carcinoma in situ of uterine cervix).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Overall Survival（OS) | 24 months
  Overall survival (OS) was defined as the time from date of randomization to date of death due to any cause.The date the patient was recorded alive of last follow-up.Median time results from unstratified Kaplan-Meier estimates.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 24 months
  PFS is defined as time from randomisation to disease progression or death whichever occurs first. Assessed by central independent review according to the Response Evaluation Criteria in Solid Tumours (RECIST 1.1).
Objective response rate (ORR) | 24 months
  ORR was defined as the proportion of patients whose best response was Complete Response [CR: disappearance of all clinical and radiological evidence of tumor (both target and non-target)] or Partial Response [PR: at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD] over the whole duration of study.
Duration of response (DoR) | 24 months
  DoR was defined as the time from documentation of tumor response to disease progression.
Disease control rate (DCR) | 24 months
  DCR was defined as the proportion of patients whose best response was CR or PR or Stable Disease (SD)
Mean Change From Baseline in European Organization for Research and Treatment of Cancer core quality of life questionnaire (EORTC QLQ-C30) | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Medical Oncology, Cancer Center, Sun Yet-sen University, Guangzhou, Guangdong
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality